CLINICAL TRIAL: NCT01419067
Title: A Phase II Trial of Limited Surgery and Proton Therapy for Craniopharyngioma and Observation for Craniopharyngioma After Radical Resection
Brief Title: A Phase II Trial of Limited Surgery and Proton Therapy for Craniopharyngioma or Observation After Radical Resection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT2CR; NCI-2011-03707 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Craniopharyngioma
Keywords: Proton Therapy; Radical resection
MeSH Terms: conditions — Craniopharyngioma | interventions — Proton Therapy; Radiotherapy; Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Craniopharyngioma Patients (Other): Craniopharyngioma patients will have limited surgery and a 5mm clinical target volume margin in combination with proton therapy. Proton therapy will be indicated for patients with diagnosed craniopharyngioma who are not treated with radical surgery (gross-total resection). Patients who have had radical surgery or limited surgery prior to enrollment on this study and have no evidence of tumor will be observed for 5 years.
  Participants receive ^1^8F-fluorodeoxyglucose and ^1^1C-methionine will be given to aid in tumor visualization.
  Interventions: Procedure: Radical Surgery or Limited Surgery; Device: Proton Therapy; Drug: ^1^8F-fluorodeoxyglucose; Drug: ^1^1C-methionine

INTERVENTIONS:
Procedure: Radical Surgery or Limited Surgery — Patients will be selected for radical surgery based on the neurosurgeon's assessment that a Gross-Total Resection may be achieved with acceptable post-operative morbidity. The goal of surgical intervention in this study should be to facilitate tumor control, keeping surgical morbidity to a minimum. Common indications for surgical intervention directed at the tumor will include establishing a tissue diagnosis, tumor control by radical resection, relieving tumor mass effect to reduce symptoms and decreasing the target volume for proton therapy by planned volume reduction surgery. These indications can be achieved through radical or limited surgery.
Device: Proton Therapy — Proton therapy will be started once a final treatment plan has been developed and approved. There is no time limit for the interval from enrollment to when proton therapy commences. The total prescribed dose will be 54CGE administered at 1.8CGE per fraction. The time course of administration will be one fraction per day, 5 days per week, for a period of 6 weeks. Radiation will be prescribed to the planning target volume which will include the tumor bed encompassed by an anatomically defined margin meant to include subclinical microscopic disease, and an additional geometric margin that is meant to account for the technical limitations associated with planning and administering daily fractionated treatment. Making radiation therapy safer through the use of proton therapy.
  Other Names: Radiation
Drug: ^1^8F-fluorodeoxyglucose — This is a contrast media that will be given intravenously to aid in tumor visualization.
  Other Names: ^1^8F-FDG; Contrast Media
Drug: ^1^1C-methionine — This is a contrast media that will be given intravenously to aid in tumor visualization.
  Other Names: Contrast Media

SUMMARY:
The goal of this study is to determine the feasibility and safety of treating patients with a brain tumor known as craniopharyngioma with limited surgery and a 5mm clinical target volume margin in combination with proton therapy. Proton therapy will be indicated for patients with diagnosed craniopharyngioma who are not treated with radical surgery (gross-total resection). Irradiated patients will undergo a series of evaluations designed to evaluate the effects of proton therapy. Similar evaluations will be performed on patients treated with radical surgery. Proton therapy will include 30 treatment fractions administered 5 days per week. Weekly imaging will be a requirement to monitor for cyst expansion and target volume deformation.

DETAILED DESCRIPTION:
The primary objectives of this study :

To estimate the progression-free and overall survival distributions for children and young adults with craniopharyngioma treated with limited surgery and proton therapy using a 5mm clinical target volume margin while monitoring for excessive central nervous system necrosis.

The Secondary Objectives of this study:

* To estimate the cumulative incidence of cystic intervention and the event-free survival distribution for children and young adults with craniopharyngioma treated with limited surgery and proton therapy using a 5mm clinical target volume margin; and compare the distributions of progression-free, event-free and overall survival with the distributions for the St. Jude Children's Research Hospital cohort of 93 patients on which the design of this trial is based.
* To estimate the distributions of progression-free survival and overall survival for children and young adults with craniopharyngioma treated only with primary surgical resection and to compare these distributions with the distributions observed for patients treated with limited surgery and proton therapy.

ELIGIBILITY:
Inclusion Criteria:

* Craniopharyngioma diagnosed by histology, cytology or neuroimaging.
* Patients ages 0-21 years at the time of diagnosis.

Exclusion Criteria

* Prior history of fractionated radiation therapy.
* Prior treatment with intracystic P-32, intracystic bleomycin or radiosurgery.
* Pregnant females are excluded. Radiation has teratogenic or abortifacient effects.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2011-08-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Estimate the progression-free and overall survival distributions for children and young adults with craniopharyngioma treated with limited surgery and proton therapy | 5 years
  Reducing the clinical target volume margin to 5mm and using proton therapy, with the goal of reducing side effects from irradiation, will not increase the rate of tumor progression compared to photon therapy with a similar or larger clinical target volume margin.

SECONDARY OUTCOMES:
Estimate the cumulative incidence of cystic intervention and the event-free survival distribution for children and young adults with craniopharyngioma treated with limited surgery and proton therapy | 5 years
  This will be improved by models based on clinical and treatment factors and longitudinal measures of CNS effects.
Estimate the distributions of progression-free survival and overall survival for children and young adults with craniopharyngioma treated only with primary surgical resection | 5 years
  This will be improved by models based on clinical and treatment factors and longitudinal measures of CNS effects

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Merchant, DO, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - University of Florida Health Proton Therapy Institute, Jacksonville, Florida
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- [Derived] Merchant TE, Hoehn ME, Khan RB, Sabin ND, Klimo P, Boop FA, Wu S, Li Y, Burghen EA, Jurbergs N, Sandler ES, Aldana PR, Indelicato DJ, Conklin HM. Proton therapy and limited surgery for paediatric and adolescent patients with craniopharyngioma (RT2CR): a single-arm, phase 2 study. Lancet Oncol. 2023 May;24(5):523-534. doi: 10.1016/S1470-2045(23)00146-8. Epub 2023 Apr 18. PMID 37084748
- [Derived] Wilson LJ, Pirlepesov F, Moskvin V, Li Z, Guo Y, Li Y, Merchant TE, Faught AM. Proton therapy delivery method affects dose-averaged linear energy transfer in patients. Phys Med Biol. 2021 Apr 1;66(7). doi: 10.1088/1361-6560/abe835. PMID 33607632
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols